CLINICAL TRIAL: NCT00772876
Title: An Open Label, Multicenter Phase I Study Of Selective Cyclin Dependent Kinase Inhibitor P1446A-05 In Subjects With Advanced Refractory Malignancies
Brief Title: A Multicenter Phase I Clinical Study of a New Compound P1446A-05 in Patients With Advanced Refractory Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Piramal Enterprises Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P1446A-05/20/08
Record Dates: First submitted 2008-10-13; First posted 2008-10-15 (Estimated); Last update posted 2012-11-22 (Estimated); Status verified 2012-11

CONDITIONS: Cancer
Keywords: P1446A-05; Advanced refractory malignancies; Phase I
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- P1446A-05 (Experimental): Single arm of the study drug. This being a dose escalation study, patient will receive a dose depending on the stage of the trial.
  Interventions: Drug: P1446A-05

INTERVENTIONS:
Drug: P1446A-05 — P1446A-05 capsules will be given once daily for 28 days in each 28 day cycle for 4 such cycles. The starting dose, for first cohort will be 75 mg once daily. Subsequent cohorts of patients will receive higher doses till the recommended phase II dose is identified.

SUMMARY:
This is a phase I study of a novel compound P1446A-05. Aim of this study is to identify the the recommended phase II dose of the drug and to determine the nature of adverse effects associated with the drug. P1446A-05 capsules will be given continuously (28 days in each 28 day cycle) to patients suffering from advanced malignancies with no effective treatment available. The dose of the study agent will be lower i.e. 75 mg per day for initial patients. If this dose is found safe, higher dose will be administered to next set of (three to six) patients. This will continued till the safest and best dose is identified. Treatment will be given for 4 cycles and continued further if found effective. Dose schedule may be modified to introduce treatment holiday,if frequent adverse effects are seen on continuous administration.

ELIGIBILITY:
Inclusion Criteria:

* Histologically and/ or cytologically confirmed solid malignant tumor or Malignant Lymphoma (excluding CNS Lymphoma and multiple myeloma) that is refractory to currently available treatment or for which no standard treatment exists
* Measurable disease
* Must have completed any prior chemotherapy, radiotherapy, biologic/targeted anti-cancer therapy or surgery at least 4 weeks (at least 6 weeks for nitrosureas and mitomycin C; 3 months for monoclonal antibodies, radioactive monoclonal antibodies or any radio- or toxin- immunoconjugates) before study entry and subjects must have recovered (to ≤grade 1) from the toxic effects from any prior therapy.
* Must not have had more than 40% of their bone marrow radiated and must have either measurable disease outside the field or progression post radiation therapy.
* Age ≥ 18 years
* ECOG performance status ≤ 2
* Life expectancy of at least 12 weeks
* Normal organ and marrow function as defined below:

Hemoglobin >/= 90 g/L Leukocytes >/=3 x 109/L Absolute Neutrophil Count (ANC) >/=1.5 x 109/L Platelets >/=100 x 109/L Total bilirubin </= 1.5 X institutional Upper Limit of Normal (ULN) AST(SGOT) </=2.5 X institutional ULN ALT(SGPT) </=2.5 X institutional ULN Creatinine </=1.5 X institutional ULN

- Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

* autologous or allogeneic bone marrow transplant within 6 months of day 1 of study drug administration
* Known brain metastases at the time of screening
* Any other investigational drug within 1 month prior to day 1 of study drug administration or not recovered (to ≤grade 1) from adverse effects of the investigational agent received prior to this period.
* History of allergic reactions attributed to compounds of similar chemical structure to P1446A-05.
* On immunosuppressive therapy.
* History of unstable angina or myocardial infarction or stroke within 6 months prior to Day 1 of study drug administration.
* Uncontrolled inter-current illness including, but not limited to active infection, symptomatic congestive heart failure, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Known to be suffering from infection with HIV, Tuberculosis, Hepatitis C or Hepatitis B.
* Pregnant or lactating women
* Women of childbearing potential [defined as a sexually mature woman who has not undergone hysterectomy or who has not been naturally postmenopausal for at least 24 consecutive months (i.e. who has had menses any time in the preceding 24 consecutive months)] and men, not agreeing to use adequate contraception (two methods of contraception, including at least one barrier method, - i.e. : hormonal and a barrier method of birth control or abstinence) prior to study entry (after signing the informed consent document), during the duration of study participation and for at least 4 weeks after withdrawal from the study drug, unless they are surgically sterilised.
* Any condition, including laboratory abnormalities, that in the opinion of the investigator places the subject at an unacceptable risk or deems the subject not suitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2008-12; Primary Completion 2012-04 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Number of Dose Limiting Toxicities at a dose level | Cycle 1 of each subject

SECONDARY OUTCOMES:
Response rate | At the end of every 2 cycles

CONTACTS AND LOCATIONS:
Overall Officials: Siu-Chung Q Chu, MD, FRCP(C), Principal Investigator — Staff Medical Oncologist, Cross Cancer Institute, Department of Medical Oncology, Edmonton, AB; Christian K Kollmannsberger, MD, Principal Investigator — Medical Oncologist, Division Medical Oncology, British Columbia Cancer Agency (BCCA), Vancouver, BC; S Welch, Principal Investigator — London Health Sciences Centre (LHSC), London, Ontario; Dr. Patricia Tang, Principal Investigator — Tom Baker Cancer Centre, Calgary, Alberta
Locations (4):
- Canada (4):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute (CCI),, Edmonton, Alberta
  - British Columbia Cancer Agency (BCCA),, Vancouver, British Columbia
  - London Health Sciences Centre (LHSC), London, Ontario

REFERENCES:
- [Derived] Malumbres M, Barbacid M. Cell cycle, CDKs and cancer: a changing paradigm. Nat Rev Cancer. 2009 Mar;9(3):153-66. doi: 10.1038/nrc2602. PMID 19238148